CLINICAL TRIAL: NCT04001634
Title: Dual Anti-HER2 Therapy (Lapatinib and Trastuzumab) Plus Chemotherapy in Metastatic HER2-positive Breast Cancer Patients- a Multicenter Retrospective Study
Brief Title: Dual Anti-HER2 Therapy (Lapatinib and Trastuzumab) Plus Chemotherapy in HER2-positive MBC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-8
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dual anti-HER2 group: Dual anti-HER2 therapy (lapatinib and trastuzumab) plus chemotherapy

SUMMARY:
To explore the real world situation of trastuzumab and lapatinib combined chemotherapy in China, and to explore the relationship between progression free survival and treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. woman, age > 18 years old 2. Diagnosed with HER2 +Metastatic Breast Cancer 3. Dual anti-HER2 therapy (lapatinib and trastuzumab) plus chemotherapy for at least one cycle, starting from 2013.09.01-2019.07.31 4. Available medical history

Exclusion Criteria:

* 1. Incomplete medical history

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival
OS | 6 weeks
  Overall survival
ORR | 6 weeks
  Objective Response Rate

SECONDARY OUTCOMES:
Treatment Pattern | 6 weeks
  Choice of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Biyun Wang, MD, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Gong C, Lu Q, Zhou Z, Luo T, Li W, Li G, Ge R, Xu F, Wang B. Real-World Data of Triplet Combination of Trastuzumab, Lapatinib, and Chemotherapy in HER2-Positive Metastatic Breast Cancer: A Multicenter Retrospective Study. Front Oncol. 2020 Mar 3;10:271. doi: 10.3389/fonc.2020.00271. eCollection 2020. PMID 32195186